CLINICAL TRIAL: NCT02839408
Title: Efficacy of Oral Probiotic and Antibiotic Administration in Clinical, Immunological and Microbiological Parameters of Patients With Chronic Periodontitis Treated With Non Surgical Periodontal Treatment
Brief Title: Efficacy of Oral Probiotic and Antibiotic Administration in Patients With Chronic Periodontitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Jorge Gamonal, Prof, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FONDECYT 1130570.b
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Periodontitis
Keywords: periodontitis; azithromycin; probiotic
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Azithromycin; Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Periodontal treatment, talc powder tab (Placebo Comparator): Periodontal treatment (scaling and root planning) and one tablet containing talc powder per day during 3 months
  Interventions: Other: Talc powder; Procedure: Periodontal treatment Scaling and root planning
- Periodontal treatment, Probitic (Experimental): Periodontal treatment (scaling and root planning) and one sachet containing Lactobacillus rhamnosus SP1 per day during 3 months.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus SP1; Procedure: Periodontal treatment Scaling and root planning
- Periodontal treatment, Antibiotic (Experimental): Periodontal treatment (scaling and root planning) and one tablet containing 500mg Azithromycin
  Interventions: Drug: Azithromycin; Procedure: Periodontal treatment Scaling and root planning

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus SP1 — Sachet containing Lactobacillus rhamnosus SP1
  Arms: Periodontal treatment, Probitic
Drug: Azithromycin — Tablet containing 500mg Azithromicyn
  Arms: Periodontal treatment, Antibiotic
Other: Talc powder — Sachet containing talc powder and tablet containing talc powder
  Arms: Periodontal treatment, talc powder tab
Procedure: Periodontal treatment Scaling and root planning

SUMMARY:
The aim of this randomized placebo- controlled clinical trial is to evaluate the effects of Lactobacillus rhamnosus SP1- containing probiotic tablets and azithromycin tablets as an adjunct to scaling and root planning (SRP).

Material and methods: Fifty-four chronic periodontitis patients will be recruited and monitored clinically, immunologically and microbiologically at baseline, 3, 6, 9 and 12 months after therapy. All patients will receive scaling and root planning and randomly will be assigned over an probiotic experimental (SRP + probiotic, n=18), antibiotic experimental (SRP + Azithromycin, n=18) or control (SRP + placebo, n=18) group. Probiotic will be used once per day during 3 months. Antibiotic will be used once per day during 5 days.

ELIGIBILITY:
Inclusion Criteria:

* 14 natural teeth, excluding third molars
* 10 posterior teeth
* 35 years old
* 5 teeth with periodontal sites with probing depths ≥5mm, clinical attachment loss ≥3mm Bleeding on probing ≥20% of sites Extensive bone loss determined radiographically

Exclusion Criteria:

* Periodontal treatment before the time of examination
* Systemic illness
* Pregnancy Anticoagulant, antibiotics and non- steroid anti- inflammatory therapy in the 6-month period before the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Differences of at least 1mm between groups for clinical attachment level changes | baseline, 3, 6, 9 and 12 month

SECONDARY OUTCOMES:
Differences between groups for probing depth changes | baseline, 3, 6, 9 and 12 month
Differences between groups for bleeding on probing changes | baseline, 3, 6, 9 and 12 month
Differences between groups for plaque index changes | baseline, 3, 6, 9 and 12 month
Differences between groups for levels of Interleukin (IL)-17, IL-8, beta-defensing 3 changes in gingival crevicular fluid | baseline, 3, 6, 9 and 12 month
Differences between groups for levels of periodontal pathogens changes | baseline, 3, 6, 9 and 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry of University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morales A, Contador R, Bravo J, Carvajal P, Silva N, Strauss FJ, Gamonal J. Clinical effects of probiotic or azithromycin as an adjunct to scaling and root planning in the treatment of stage III periodontitis: a pilot randomized controlled clinical trial. BMC Oral Health. 2021 Jan 7;21(1):12. doi: 10.1186/s12903-020-01276-3. PMID 33413320